CLINICAL TRIAL: NCT02678000
Title: A Two Part Randomized, Double-blind, Parallel-group, Placebo-controlled Study to Evaluate the Renal Safety, Tolerability and Pharmacokinetics of LHW090 in Patients With Moderately Impaired Renal Function on Angiotensin Receptor Blockers
Brief Title: Study of the Safety, Tolerability, and Pharmacokinetics of LHW090 in Patients With Moderately Impaired Renal Function
Acronym: LHW090
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLHW090X2102
Record Dates: First submitted 2016-01-29; First posted 2016-02-09 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Chronic Kidney Disease (CKD)
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LHW090 (Experimental): For Part 1, patients will receive 3 doses of LHW090 once daily with escalating doses every 4 days for a total 12 days of treatment.
  For Part 2, patients will receive LHW090 once daily for 4 weeks.
  Interventions: Drug: LHW090
- Placebo (Placebo Comparator): For Part 1, patients will receive matching placebo once daily for 12 days. For Part 2, patients will receive matching placebo once daily for 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LHW090 — LHW090 is orally administered
  Arms: LHW090
Drug: Placebo — Matching placebo of LHW090
  Arms: Placebo

SUMMARY:
This was a randomized, double-blind, parallel group, placebo-controlled study, in two sequential parts that evaluated the renal safety, tolerability and pharmacokinetics of LHW090 in patients with moderately impaired renal function.

ELIGIBILITY:
Inclusion Criteria (all Parts):

* Written informed consent must be obtained before any assessment is performed.
* Male and female patients, age 40 to 85 years of age (inclusive) on a stable (at least 1 month) dose of an angiotensin receptor blocker (ARB) and stable moderately impaired renal function, defined here as an eGFR 30-59 mL/min/1.73m^2 (inclusive) using the 4 variable MDRD Study equation for at least 3 months.
* At screening, vital signs (systolic and diastolic blood pressure and pulse rate) will be assessed in the sitting position after the patient has rested for at least five minutes, and again after three minutes in the standing position. Sitting vital signs should be within the following ranges:

  * oral body temperature between 35.0-37.5 °C
  * systolic blood pressure, 100-170 mm Hg
  * diastolic blood pressure, 50-100 mm Hg
  * pulse rate, 50 - 95 bpm
* Patients should be excluded if their standing vital signs (relative to sitting) show findings which, in the opinion of the Investigator, are associated with clinical manifestation of postural hypotension (i.e. absence of any other cause). The Investigator should carefully consider enrolling patients with either a > 20 mm Hg decrease in systolic or a >10 mm Hg decrease in diastolic blood pressure, accompanied by a > 20 bpm increase in heart-rate (comparing standing to sitting results).
* Patients must weigh at least 50 kg to participate in the study, and must have a body mass index (BMI) within the range of 18 - 38 kg/m^2. BMI = Body weight (kg) / [Height (m)]^2.
* Able to communicate well with the investigator, to understand and comply with the requirements of the study.

Exclusion criteria:

* History of angioedema, drug-related or otherwise, as reported by the patient.
* Use of angiotensin converting enzyme inhibitors (ACE inhibitors), mineralocorticoid receptor antagonists (e.g. spironolactone or eplerenone), aliskiren, vasopressin receptor antagonists (e.g. tolvaptan), or oral alkalinizing agents (e.g. sodium and potassium citrate or Shohl's solution). Note: Patients who discontinue their ACE-inhibitor and substitute with an angiotensin receptor blocker (ARB) may be eligible to be rescreened provided their medication regimen has been stable for at least 1 month and their renal function has been stable for at least 3 months. Any substitutions or changes to a patient's medication regimen must be done under the guidance of the patient's treating physician.
* History of a renal transplant.
* Known current significant left ventricular outflow obstruction, such as obstructive hypertrophic cardiomyopathy or significant severe valvular disease on prior or current echocardiogram.
* A serum potassium ≤ 3.5 mmol/l or ≥ 5.2 mmol/l at screening.
* A previous history or previously diagnosed renal cystic disease such as autosomal dominant polycystic kidney disease (history of an incidental asymptomatic acquired renal cyst(s) is excepted); obstructive uropathy; renal stone(s) in the past 2 years; chronic interstitial nephropathy; drug induced nephropathy; residual renal insufficiency following an episode of acute kidney injury or acute tubular necrosis related to renal atheroembolic disease, septic shock or ischemic nephropathy; renal tubular acidosis requiring treatment; nephrotic syndrome or nephrotic range proteinuria; or renal artery stenosis.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2018-10-11 (Actual); Study Completion 2018-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (12):
- United States (7):
  - Novartis Investigative Site, Anaheim, California
  - Novartis Investigative Site, Lakewood, Colorado
  - Novartis Investigative Site, Miami Lakes, Florida
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, New Orleans, Louisiana
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Saint Paul, Minnesota
- Germany (5):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Elsterwerda
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Mannheim

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=310

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects (N=11) who enrolled in in PART 1 completed the study : LHW090 (N=7) and placebo (N=4). Of all subjects (N=73) in PART 2, a total of 69 subjects completed and 4 subjects discontinued.
Pre-assignment Details: All subjects (N=11) who enrolled in in PART 1 completed the study : LHW090 (N=7) and placebo (N=4). Of all subjects (N=73) in PART 2, a total of 69 subjects completed and 4 subjects discontinued.
Groups:
- LHW090 (PART 1): For Part 1, patients will receive 3 doses of LHW090 once daily with escalating doses every 4 days for a total 12 days of treatment.
- Placebo (PART 1): For Part 1, patients will receive matching placebo once daily for 12 days.
- LHW090 100mg (PART 2): For PART 2, patients will receive LWH090 100 mg for 4 weeks
- LHW090 200mg (PART 2): For PART 2, patients will receive LWH090 200 mg for 4 weeks
- Placebo (PART 2): For Part 2, patients will receive matching placebo once daily for 4 weeks.
Period: PART 1
Arm/Group | LHW090 (PART 1) | Placebo (PART 1) | LHW090 100mg (PART 2) | LHW090 200mg (PART 2) | Placebo (PART 2)
Started | 7 | 4 | 0 | 0 | 0
Completed | 7 | 4 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: PART 2
Arm/Group | LHW090 (PART 1) | Placebo (PART 1) | LHW090 100mg (PART 2) | LHW090 200mg (PART 2) | Placebo (PART 2)
Started | 0 | 0 | 28 | 27 | 18
Completed | 0 | 0 | 25 | 26 | 18
Not Completed | 0 | 0 | 3 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LHW090 (PART 1) | Placebo (PART 1) | LHW090 100mg (PART 2) | LHW090 200mg (PART 2) | Placebo (PART 2) | Total
Number analyzed (Participants) | 7 | 4 | 28 | 27 | 18 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.3 (3.64) | 67.5 (16.01) | 71.0 (9.18) | 69.0 (8.82) | 65.3 (11.58) | 68.8 (9.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 8 | 10 | 9 | 31
  Male | 6 | 1 | 20 | 17 | 9 | 53
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 3 | 0 | 6
  White | 6 | 3 | 27 | 24 | 18 | 78
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Reported Adverse Events Receiving Escalating Doses of LHW090 (Part 1)
Description: Any sign or symptom that occurs during the study treatment plus the 30 days post treatment. For LHW090, incidence of AEs by primary organ class presented
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment, (12 days dosing period + 9 days follow up (PART 1) plus 30 days post treatment, up to maximum duration of approximately 20 months
Population: Safety Analysis Set -All subjects that received study drug and with no protocol deviations with relevant impact on safety
Measure: Number; unit: Count of Participants
Groups:
- LHW090 25 mg (PART 1): For Part 1, patients will receive 3 doses of LHW090 25 mg once daily with escalating doses every 4 days for a total 12 days of treatment.
- LHW090 50 mg (PART 1): For Part 1, patients will receive 3 doses of LHW090 50 mg once daily with escalating doses every 4 days for a total 12 days of treatment.
- LHW090 100 mg (PART 1): For Part 1, patients will receive 3 doses of LHW090 100 mg once daily with escalating doses every 4 days for a total 12 days of treatment.
Arm/Group | LHW090 25 mg (PART 1) | LHW090 50 mg (PART 1) | LHW090 100 mg (PART 1) | Placebo (PART 1)
Number analyzed (Participants) | 7 | 7 | 7 | 4
Count of Participants
  Number of patients with at least one AE | 1 | 0 | 1 | 2
  Gastrointestinal disorders | 1 | 0 | 1 | 2
  Skin and subcutaneous tissue disorders | 0 | 0 | 1 | 2
  General disorders & administration site conditions | 0 | 0 | 0 | 1
  Musculoskeletal and connective tissue disorders | 0 | 0 | 0 | 1
  Nervous system disorders | 0 | 0 | 0 | 1
  Psychiatric disorders | 0 | 0 | 0 | 1

2. Primary Outcome: Pharmacokinetics of LHW090/LHV527 (Active Metabolite) in Plasma: Area Under the Plasma Concentration-time Curve From Time Zero Time 't' Where t is a Defined Time Point After Administration (AUC0-t) (PART 1)
Description: The area under the plasma concentration-time curve from time zero to 24 hours. Area Under the Curve (AUC0-t) after 4 days dosing will be reported for PART 1. LHW090 and LHV527 (its active metabolite)
Time Frame: Within 60 minutes prior to dosing, post dose +/- 10 min from greater or equal to 1 hr to 24 hrs.
Population: PK Analysis Set -Subjects with at least one available valid PK concentration measurement, who received study drug and experienced no protocol deviations with relevant impact on PK data
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- LHW090/LHV527 25 mg (PART 1): For Part 1, patients will receive 3 doses of LHW090 25 mg once daily with escalating doses every 4 days for a total 12 days of treatment. (PK draw with active metabolite, LHV527)
- LHW090/LHV527 50 mg (PART 1): For Part 1, patients will receive 3 doses of LHW090 50 mg once daily with escalating doses every 4 days for a total 12 days of treatment. (PK draw with active metabolite, LHV527)
- LHW090/LHV527 100 mg (PART 1): For Part 1, patients will receive 3 doses of LHW090 100 mg once daily with escalating doses every 4 days for a total 12 days of treatment. (PK draw with active metabolite, LHV527)
Arm/Group | LHW090 25 mg (PART 1) | LHW090 50 mg (PART 1) | LHW090 100 mg (PART 1) | LHW090/LHV527 25 mg (PART 1) | LHW090/LHV527 50 mg (PART 1) | LHW090/LHV527 100 mg (PART 1)
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 7 | 7
h*ng/mL | 3750 (815) | 7150 (1480) | 13900 (2180) | 19200 (3990) | 36500 (5720) | 68800 (11800)

3. Primary Outcome: Number of Patients Who Developed a Renal Event (PART 2)
Description: Patients who developed a renal event will be reported (defined as a ≥0.3 mg/dL increase in serum creatinine from baseline within 24-48 hours post dose )
Time Frame: Baseline, within 24 to 48 hours of post-dose weekly for up to 8 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- LHW090 100mg (PART 2): For PART 2, patients will receive LWH090 100 mg once daily for 4 weeks
- LHW090 200mg (PART 2): For PART 2, patients will receive LWH090 200 mg once daily for 4 weeks
Arm/Group | LHW090 100mg (PART 2) | LHW090 200mg (PART 2) | Placebo (PART 2)
Number analyzed (Participants) | 28 | 27 | 18
Participants | 0 | 1 | 0

4. Secondary Outcome: Cmax : Pharmacokinetics of LHW090/LHV527 (Active Metabolite) in Plasma: Observed Maximum Plasma Concentration Following Administration of LHW090 (PART 1/PART 2)
Description: The observed maximum plasma (or serum or blood) concentration following drug administration for PART 1 and PART 2
Time Frame: PART 1: within 60 minutes prior to dosing, post dose +/- 10 min from greater or equal to 1 hr to 24 hrs. PART 2: within 60 min +/- 10 min from greater or equal to 1 hr to 8 hours after 4 weeks dosing.
Population: PK Analysis Set - Subjects with at least one available valid PK concentration measurement, who received study drug and experienced no protocol deviations with relevant impact on PK data
Measure: Mean (Standard Deviation); unit: ng / mL
Arm/Group | LHW090 25 mg (PART 1) | LHW090 50 mg (PART 1) | LHW090 100 mg (PART 1) | LHW090 100mg (PART 2) | LHW090 200mg (PART 2)
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 7
ng / mL
  PK Value for LHW090: number analyzed (Participants) | 7 | 7 | 7 | 6 | 6
  PK Value for LHW090 | 1160 (589) | 2000 (1020) | 4230 (1400) | 4470 (1690) | 7530 (3750)
  PK Value for LHW090/LHV527(active metabolite): number analyzed (Participants) | 6 | 7 | 7 | 6 | 6
  PK Value for LHW090/LHV527(active metabolite) | 1690 (338) | 3070 (682) | 5100 (734) | 6200 (1560) | 10300 (1440)

5. Secondary Outcome: AUC0-t: Pharmacokinetics of LHW090/LHV527 (Active Metabolite)in Plasma: Area Under the Plasma Concentration-time Curve From Time Zero Time 't' Where t is a Defined Time Point After Administration (PART 2)
Description: The area under the plasma concentration-time curve from time zero to 24 hours
Time Frame: PART 2: within 60 min +/- 10 min from greater or equal to 1 hr to 8 hours after 4 weeks dosing
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h* ng/mL
Groups:
- LHW090 100 mg (PART 2): For PART 2, patients will receive LWH090 100 mg once daily for 4 weeks
- LHW090/LHV527 100 mg (PART 2): For PART 2, patients will receive LWH090 100 mg once daily for 4 weeks. (PK draw with active metabolite, LHV527)
- LHW090/LHV527 200 mg (PART 2): For PART 2, patients will receive LWH090 200 mg once daily for 4 weeks. (PK draw with active metabolite, LHV527)
Arm/Group | LHW090 100 mg (PART 2) | LHW090 200mg (PART 2) | LHW090/LHV527 100 mg (PART 2) | LHW090/LHV527 200 mg (PART 2)
Number analyzed (Participants) | 28 | 27 | 28 | 27
h* ng/mL | 21500 (6810) | 42900 (20700) | 96700 (32800) | 181000 (51100)

6. Secondary Outcome: Tmax: Pharmacokinetics of LHW090/LHV527 in Plasma: Time to Reach the Maximum Concentration After Administration of LHW090 (PART 1/PART 2)
Description: The time to reach the maximum concentration after drug administration
Time Frame: as for outcome 4
Population: PK Analysis Set-Subjects with at least one available valid PK concentration measurement, who received study drug and experienced no protocol deviations with relevant impact on PK data
Measure: Median (Full Range); unit: hour (hr)
Arm/Group | LHW090 25 mg (PART 1) | LHW090 50 mg (PART 1) | LHW090 100 mg (PART 1) | LHW090 100mg (PART 2) | LHW090 200mg (PART 2)
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 7
hour (hr)
  PK Value for LHW090: number analyzed (Participants) | 7 | 7 | 7 | 6 | 6
  PK Value for LHW090 | 2.00 [1.00 to 3.00] | 1.02 [1.00 to 3.00] | 1.00 [1.00 to 4.00] | 2.00 [1.00 to 4.00] | 2.50 [1.00 to 12.0]
  PK Value for LHW090/LHV527(active metabolite): number analyzed (Participants) | 6 | 7 | 7 | 6 | 6
  PK Value for LHW090/LHV527(active metabolite) | 3.58 [2.00 to 12.0] | 4.00 [2.00 to 12.0] | 4.00 [2.00 to 8.00] | 3.00 [2.00 to 8.00] | 4.00 [3.00 to 12.0]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment, plus 30 days post treatment, up to maximum duration of approximately 20 months
Description: Any sign or symptom that occurs during the study treatment plus the 30 days post treatment.
Groups:
- PART 1 Placebo: For Part 1, patients will receive matching placebo once daily for 12 days.
- LHW090 200 mg (PART 2): For PART 2, patients will receive LWH090 200 mg once daily for 4 weeks
- Placebo (PART 2: For Part 2, patients will receive matching placebo once daily for 4 weeks.
Arm/Group | LHW090 25 mg (PART 1) | LHW090 50 mg (PART 1) | LHW090 100 mg (PART 1) | PART 1 Placebo | LHW090 100mg (PART 2) | LHW090 200 mg (PART 2) | Placebo (PART 2
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7 | 0/7 | 0/4 | 0/28 | 0/27 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/7 | 0/4 | 3/28 | 0/27 | 0/18
Other Adverse Events (participants affected / at risk) | 1/7 | 0/7 | 1/7 | 2/4 | 13/28 | 16/27 | 9/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LHW090 25 mg (PART 1) (N=7) | LHW090 50 mg (PART 1) (N=7) | LHW090 100 mg (PART 1) (N=7) | PART 1 Placebo (N=4) | LHW090 100mg (PART 2) (N=28) | LHW090 200 mg (PART 2) (N=27) | Placebo (PART 2 (N=18)
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LHW090 25 mg (PART 1) (N=7) | LHW090 50 mg (PART 1) (N=7) | LHW090 100 mg (PART 1) (N=7) | PART 1 Placebo (N=4) | LHW090 100mg (PART 2) (N=28) | LHW090 200 mg (PART 2) (N=27) | Placebo (PART 2 (N=18)
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2 | 4 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0
Infusion site haemorrhage (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Xerosis (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Blood pressure decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Lactose intolerance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Apathy (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasal pruritus (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 6 | 1 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-08-07): https://cdn.clinicaltrials.gov/large-docs/00/NCT02678000/Prot_001.pdf
  • Statistical Analysis Plan (2018-12-21): https://cdn.clinicaltrials.gov/large-docs/00/NCT02678000/SAP_000.pdf